CLINICAL TRIAL: NCT03259282
Title: Gammaglobulins Level is Predictive Factor of Evolution in Sarcoidosis
Acronym: GAMES
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC16_3046_GAMES
Record Dates: First submitted 2017-08-21; First posted 2017-08-23 (Actual); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Sarcoidosis
MeSH Terms: conditions — Sarcoidosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Analysis of gamma globulin — Electrophoresis of proteins

SUMMARY:
Evaluation of the rate of achievement of serum protein electrophoresis (PPE) in diagnosis in a retrospective cohort of patients at Rennes University Hospital

DETAILED DESCRIPTION:
In 50% of cases, sarcoidosis is associated with polyclonal hypergammaglobulinemia. The other forms have a normal gamma globulin level.

The level of gamma globulinemia has not yet been studied as an evolutionary predictive factor. Furthermore, there are disseminated granulomatoses sharing common characteristics with sarcoidosis, associated with Common Variable Immunodeficiency deficit (DICV) type Primary Immunodeficiency syndrome (DIP), thus occurring in hypogammaglobulinemic patients.

ELIGIBILITY:
Inclusion Criteria:

- Patients newly diagnosed with sarcoidosis

Exclusion Criteria:

* Comorbidity responsible for a change in the level of gamma globulin
* Other etiology of granulomatosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with sarcoidosis
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2017-03-07 (Actual); Primary Completion 2017-03-22 (Actual); Study Completion 2017-03-22 (Actual)

PRIMARY OUTCOMES:
Study of gamma globulin level present in the blood at the time of diagnosis of sarcoidosis on disease activity | Day 1
  Electrophoresis rates of serum proteins
Study of gamma globulin level present in the blood at the time of diagnosis of sarcoidosis on the course of the disease | Day 1
  Electrophoresis rates of serum proteins

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Rennes, Rennes, France

IPD SHARING:
Plan to Share IPD: No